CLINICAL TRIAL: NCT03883867
Title: Vaginal Tactile Imaging in Assessment of Pelvic Floor Conditions Before the Delivery
Status: Completed | Type: Observational
Sponsor: Advanced Tactile Imaging, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VTI 10
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Pelvic Floor; Perineal Rupture; Obstetric Trauma
Keywords: Pelvic Floor, Perineal Rapture, Obstetric Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Normal: The subject population will involve 10 non-pregnant women. The tactile imaging reprifucibility sub-group will include 5 non-pregnant subjects with 2 tactile imaging examinations completed in one session. All other subjects will have a single tactile imaging examination.
- Pregnant: The subject population will involve 10 pregnant women without known complications at 36-37 weeks of pregnancy scheduled for a regular examination. All pregnant subjects should be examined weekly after completing 36th week of an uncomplicated pregnancy. Routine gynecologic examination includes external and internal obstetrical examination.

SUMMARY:
The mechanical demands placed on the pelvic floor structures during vaginal delivery often exceed physiological tissue limits, resulting in maternal childbirth trauma, considerable postpartum morbidity, and increased risk of pelvic floor disorders(PFD). Injury to the perineum, vaginal supportive tissues, and pelvic floor muscles cause pain, infection, and dyspareunia, as well as pelvic organ prolapse(POP).Pregnancy and vaginal delivery are considered as a main risk factors in weakening the pelvic floor support and development of SUI, AI, and POP. CS is not only available countermeasure to reduce occurrence of obstetric trauma. Tactile imaging allows acquisition of 3D stress-strain data and 3D elasticity imaging or soft tissues.

DETAILED DESCRIPTION:
The long - term of this project is to develop, validate, and integrate into clinical practice a new paradigm and a novel device to simultaneously measure the biomechanical properties of various pelvic structural components that are impacted during vaginal delivery, and to develop a risk prediction model of maternal birth injury. Ultimately, such a model will enable individualized patient counseling regarding the mode of delivery and/or the need for obstetrical interventions to reduce child birth trauma. The approach will utilize the vaginal tactile imaging technology that the investigators have developed and validated for clinical use.

The benefits to physicians, patients and society are expected to be significant because the painful event in woman's life , given the large proportion of women suffer PFD caused by childbirth.

This new system may open a new technical capability in woman's healthcare and change the established clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women (Princeton Urogynecology, Princeton, NJ)
* Pregnant women after completed 35th week of pregnancy with fetus in vertex position and premise of vaginal delivery (Division of Maternal-Fetal Medicine, Rutgers Robert Wood Johnson Medical School, New Brunswick, NJ)

Exclusion Criteria:

* Prior perineal surgery
* HIV or hepatitis B positive serology
* Warty lesions on the vulva
* Extensive varicose veins on the vulva
* Aactive skin infection or ulceration within the vagina/vulva
* Presence of vaginal septum
* Severe hemorrhoids
* Stillbirth or extensive congenital abnormalities of the fetus

Min Age: 21 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — women in reproductive age
Study Population: The subject population will include 20 subjects. First group involves 10 non-pregnant women 5 of them will have 2 tactile imaging examinations completed in one session 5 others will have single tactile imaging examination.
  Second group involves 10 pregnant women without known complications at 36-37 weeks of pregnancy scheduled for a regular examination. All pregnant subjects should be examined weekly after completing 36 week of an uncomplicated pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Prineum elasticity | During examination procedure
  Measurement in units of elasticity, Young's modulus, kPa
Distance between pubic bone and perineum at 20 kPa load | During examination procedure
  Measurement in unit of distance, mm

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Egorov, PhD, Principal Investigator — Advanced Tactile Imaging, Inc.
Locations (3):
- United States (2):
  - Rutgers The State University Of New Jersey, New Brunswick, New Jersey
  - Princeton Urogynecology, Princeton, New Jersey
- Department of Gynecology and Obstetrics University Hospital, Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No
Will be published.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT03883867/Prot_ICF_000.pdf